CLINICAL TRIAL: NCT02356822
Title: Sarah Cannon Outcomes Registry
Status: Withdrawn | Type: Observational
Why Stopped: closed early with no results/no data collected.
Sponsor: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: SCRI HEOR_01
Record Dates: First submitted 2015-01-20; First posted 2015-02-05 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2019-06

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

INTERVENTIONS:
Other: Patient registry — Oncology data registry

SUMMARY:
This is an investigational multi-site outcomes registry intended to collect information about a patient's cancer care. Patients may enter the Registry at any time during the patient's current stage in the continuum of care. The registries main objectives will be to measure and evaluate the effects of patient care throughout the care continuum, resulting in the identification of the most effective treatment options. Objectives will encompass evaluations and analytics around safety, effectiveness, and improved efficiencies.

DETAILED DESCRIPTION:
Q

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Patients that have been diagnosed with/ or are thought to have any form of cancer at any stage in the continuum of their care from screening through survivorship.
* Patient must have the ability to understand the nature of the trial and give written informed consent

Exclusion Criteria:

* There are no exclusion criteria for this Outcomes Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18yrs or older, that have been diagnosed with/ or are thought to have any form of cancer at any stage in the continuum of their care from screening through survivorship. Patient must have the ability to understand the nature of the trial and give written informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
quality improvement | 10 yrs
Treatment patterns and utilization | 5 yrs

SECONDARY OUTCOMES:
Humanistic and economic outcomes | 10 yrs

OTHER OUTCOMES:
safety and effectiveness | 10 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Richard Geer, MD, Principal Investigator — Sarah Cannon
Locations (1):
- SCRI, Nashville, Tennessee, United States